CLINICAL TRIAL: NCT06341049
Title: Effect of Three Different Postcesarean Analgesic Techniques on ObsQoR-10 Score: Prospective, Randomized Trial
Brief Title: Effect of Three Different Postcesarean Analgesic Techniques on QbsQor-10 Score
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Aysenur Dostbil, Clinical Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-03/14
Record Dates: First submitted 2024-03-19; First posted 2024-04-02 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Recovery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Intraperitoneal local anasthetic+ loal anesthetic wound infiltration (Active Comparator): For Group Intraperitoneal local anasthetic+ loal anesthetic wound infiltration, after the birth of the newborn and placenta, the uterus is taken out and closed, the blood accumulated in the pelvis is carefully wiped with surgical towels, and after complete hemostasis is achieved, sterilely prepared 20 ml 0.5% bupivacaine + 20 ml 2% lidocaine +1 A total of 40 ml of solution containing 200,000 epinephrine will be given to the surgeon. 10 ml of this solution will be instilled into all four quadrants of the uterus before closing the parietal peritoneum or fascia. The parietal peritoneal layer will be sutured or left open, depending on the surgeon's preference. 10 ml will be infiltrated around the edges of the rectus aponeurosis, and the remaining 20 ml will be infiltrated subcutaneously into the wound area.
  Interventions: Procedure: Intraperitoneal local anasthetic application + local anesthetic wound infiltration
- Group Morphine (Active Comparator): Group Morphine will be given 11.2 mg hyperbaric bupivacaine + 15 µg fentanyl + 150 µg morphine into the spinal space.
  Interventions: Procedure: Intrathecal morphine application
- Group Quadratus lumborum block (Active Comparator): In Group Quadratus lumborum block, Quadratus lumborum block type I, a total of 40 ml of a solution containing 20 ml of 0.5% bupivacaine + 20 ml of 2% lidocaine + 1:200,000 epinephrine will be applied bilaterally under ultrasound guidance.
  Interventions: Procedure: Quadratus lumborum block tip 1 application

INTERVENTIONS:
Procedure: Intraperitoneal local anasthetic application + local anesthetic wound infiltration — For Group Intraperitoneal local anasthetic+ loal anesthetic wound infiltration, after the birth of the newborn and placenta, the uterus is taken out and closed, the blood accumulated in the pelvis is carefully wiped with surgical towels, and after complete hemostasis is achieved, sterilely prepared 20 ml 0.5% bupivacaine + 20 ml 2% lidocaine +1 A total of 40 ml of solution containing 200,000 epinephrine will be given to the surgeon. 10 ml of this solution will be instilled into all four quadrants of the uterus before closing the parietal peritoneum or fascia. The parietal peritoneal layer will be sutured or left open, depending on the surgeon's preference. 10 ml will be infiltrated around the edges of the rectus aponeurosis, and the remaining 20 ml will be infiltrated subcutaneously into the wound area.
  Arms: Group Intraperitoneal local anasthetic+ loal anesthetic wound infiltration
Procedure: Intrathecal morphine application — Group Morphine will be given 11.2 mg hyperbaric bupivacaine + 15 µg fentanyl + 150 µg morphine into the spinal space.
  Arms: Group Morphine
Procedure: Quadratus lumborum block tip 1 application — In Group Quadratus lumborum block, Quadratus lumborum block type I, a total of 40 ml of a solution containing 20 ml of 0.5% bupivacaine + 20 ml of 2% lidocaine + 1:200,000 epinephrine will be applied bilaterally under ultrasound guidance.
  Arms: Group Quadratus lumborum block

SUMMARY:
The aim of this study is to evaluate the effects of three different postsesarean analgesia techniques, including instillation of local anesthetic into the peritoneum with infiltration into all layers of the anterior abdominal wall, intrathecal morphine injection with local anesthetic, and quadrotus lumborum type 1 block, on the postoperative recovery of women using the ObsQoR-10 score..

DETAILED DESCRIPTION:
This study will be planned on women who will undergo elective cesarean section surgery with neuraxial anesthesia, after obtaining ethics committee approval and written informed consent from the patients.Parturients will be randomized by the statistician using a computerized random numbers table and divided into 3 equal groups: Group IPLA + LWI, Group QLB 1 and Group M.Postoperatively, patients' ObsQoR-10 scores will be evaluated and recorded at the 24th and 48th hours.

ELIGIBILITY:
Inclusion Criteria:

* Elective cesarean section under spinal anesthesia
* Full-term singleton pregnancy
* Agree to participate in the study
* American Society of Anaesthesiology Score of II

Exclusion Criteria:

* Contrindication for neuraxial anesthesia
* ASA≥3, diabetes, preeclampsia, cardiovascular disease, chronic pain and neuropathic pain
* Age< 18 or > 50
* Multiple pregnancy
* Presence of psychiatric diseases
* Gave a history of allergic to any medication in the study protocol
* Gave a history of chronic pain
* Unable to consent
* BMI>35 kg/m2
* Those who were given opioids during the operation due to intraoperative pain
* Those who have had previous abdominal surgery
* Patients who failed spinal anesthesia and switched to general anesthesia
* Those who have excessive bleeding or uterine atony during the operation
* Does not understand VAS
* Those who have a drain placed in the area to be infiltrated
* Gave a history of drug addiction

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Elective cesarean section patients are included in our study.
Enrollment: 120 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
obstetric quality of recovery-10 (ObsQoR-10) scores of parturient at the 24th and 48th postoperative hours | Postoperative 24th and 48th hours
  For post-cesarean analgesia, patients will receive instillation of local anesthetic into the peritoneum with infiltration into all layers of the anterior abdominal wall, intrathecal morphine injection with local anesthetic, and quadrotus lumborum type 1 block. ObsQoR-10 scores of the patients will be evaluated at the 24th and 48th hours postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Aysenur Dostbil, Study Director — Ataturk University
Locations (1):
- Ataturk University, Erzurum, Palandoken, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No